CLINICAL TRIAL: NCT06209957
Title: Evaluation of Platelet-Rich Plasma Injection vs. Corticosteroid Injection in Idiopathic Carpel Tunnel Syndrome
Brief Title: Study of Single Platelet-Rich Plasma Local Injection Vs. Single Corticosteroid Local Injection in Carpal Tunnel Syndrome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Menoufia University (Other)
Responsible Party: Principal Investigator, Aya Allam, Teaching Assistant of physical medicine, rheumatology and rehabilitation, Menoufia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PRP in CTS
Record Dates: First submitted 2023-12-27; First posted 2024-01-18 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Carpal Tunnel Syndrome
Keywords: Carpal Tunnel Syndrome; Corticosteroids; Platelet-Rich Plasma; Nerve Conduction Study; Boston Questionnaire; Visual Analogue Scale
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Intervention Model Description: A prospective, interventional, comparative double-blinded study.
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group I (Active Comparator): Local corticosteroid injection in group I: 1 ml of triamcinolone acetonide (40 milligram/1.0 mL) was locally injected in the wrist using a 25-gauge needle, which was slowly inserted 1 cm proximal to the distal wrist-flexion crease just on the radial side of the palmaris longus tendon. The injection was held if the patient experienced pain or a sensation of pins and needles in the median nerve distribution.
  Interventions: Drug: Local corticosteroid injection
- Group II (Active Comparator): Local PRP injection in group II: 2 ml of PRP was injected using the same technique of corticosteroid local injection after 2-step centrifugation of the patient's blood using a specific device. Non-steroidal anti-inflammatory drugs were avoided for two weeks before and after the procedure to prevent the possibility of inhibition of platelet function.
  Interventions: Drug: Platelet-rich Plasma Local injection

INTERVENTIONS:
Drug: Local corticosteroid injection — Local corticosteroid injection;1 ml of triamcinolone acetonide 40 milligram/1.0 mL
  Arms: Group I
Drug: Platelet-rich Plasma Local injection — Platelet-rich Plasma (From 2-step centrifugation of patient blood) Local injection.
  Arms: Group II

SUMMARY:
This clinical trial aims to evaluate the effect of a single local platelet-rich plasma injection Versus local steroid injection in treating mild idiopathic carpal tunnel syndrome regarding pain relief and function improvement and electrophysiological studies of the median nerve as a baseline and during a follow-up period of 3 months.

The main question[s] it aims to answer are:

* Does platelet-rich plasma injection provide better pain relief for CTS symptoms than steroid injection?
* Does platelet-rich plasma improve parameters of median nerve conduction study than local steroid?

Participants will have:

* A complete history and clinical examination, including sensory and motor examination and provocative tests for CTS.
* Visual analog scale (VAS), Symptom severity scale (SSS), and functional severity scale (FSS) of the Boston Carpal Tunnel Questionnaire (BCTQ) before local injection and three months after local injection by the same investigator.
* Nerve conduction studies (NCS) for median and ulnar nerves were carried out before local injection and three months after local injection by the same investigator.

Researchers will compare the efficacy of a single PRP local injection compared to a single corticosteroid local injection for treating mild idiopathic CTS using nerve conduction studies (NCS), Visual Analog Scale (VAS), and Boston Carpal Tunnel Questionnaire (BCTQ) as objective and subjective outcome measures.

DETAILED DESCRIPTION:
Carpal tunnel syndrome (CTS) is the most known entrapment neuropathy. Diagnosis of CTS is clinical, which could be confirmed by nerve conduction study (NCS). Non-operative management is the first line of treatment, including splitting, antiinflammatory, and neurotonics.

There is evidence of improvement in CTS after local corticosteroid injection, but complications are still recorded [5]. Platelet-rich plasma (PRP) is a novel, promising treatment providing growth factors for nerve regeneration and inflammation relief. This field needs further evaluation and analysis compared to traditional local steroid injection.

ELIGIBILITY:
Inclusion Criteria:

* Patients with mild primary CTS complaining of paresthesia in the palmar aspect of lateral three and half fingers of the hand. They are selected clinically and confirmed according to Padua's Neurophysiologic Severity Scale (PNSS) for CTS

Exclusion Criteria:

* Patients were excluded if they had moderate-to-severe NCS findings, space-occupying lesions within the carpal tunnel, traumatic CTS, pregnancy, diabetes mellitus, rheumatoid arthritis, or previous CTS surgery.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
Visual analog scale | before and after three months from injection time
  The pain severity was determined by the patients, on a scale of 0 (no pain) to 10 (agonizing pain)
Symptom severity scale of the Boston Carpal Tunnel Questionnaire | before and after three months from injection time
  Pain severity evaluation
Functional severity scale of the Boston Carpal Tunnel Questionnaire | before and after three months from injection time
  Hand function evaluation
Median nerve sensory peak latency | before and after three months from injection time
  Sensory conduction evaluation of median nerve
Median nerve distal motor latency | before and after three months from injection time
  Motor conduction evaluation of the median nerve.
Median nerve sensory amplitude | before and after three months from injection time
  Sensory conduction evaluation of the median nerve
Median nerve motor amplitude | before and after three months from injection time
  Motor conduction evaluation of the median nerve.
Median nerve sensory conduction velocity | before and after three months from injection time
  Sensory conduction evaluation of the median nerve
Median nerve motor conduction velocity | before and after three months from injection time
  Motor conduction evaluation of the median nerve.

CONTACTS AND LOCATIONS:
Overall Officials: Saga F El-Gazzar, Study Director — Menoufia University
Locations (1):
- Faculty of Medicine, Menoufia University, Shibīn al Kawm, Menoufia, Egypt

IPD SHARING:
Plan to Share IPD: No
Patient enrollment started June 2017 to early January 2019